CLINICAL TRIAL: NCT00655148
Title: Clinical Trial Comparing the Safety and Immunogenicity of Two Combined Diphtheria, Tetanus, Acellular Pertussis, and Inactivated Poliovirus (DTaP-IPV) Vaccines Administered to Healthy Children at 2, 3½, and 16 Months of Age
Brief Title: Safety and Immunogenicity of a New Serum-free DTaP-IPVvero Combination Vaccine
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Statens Serum Institut (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: VIPV-03
Record Dates: First submitted 2008-04-03; First posted 2008-04-09 (Estimated); Last update posted 2013-01-21 (Estimated); Status verified 2013-01

CONDITIONS: Active Immunization
Keywords: DTaP-IPV; Clinical Trial; Safety; Immunogenicity

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- A (Experimental): DTaP-IPV vero vaccination at 2, 3½, 5 and 16 months of age
  Interventions: Biological: DTaP-IPV vero vaccine
- B (Active Comparator): DTaP-IPV mkc vaccination at 2, 3½, 5 and 16 months of age
  Interventions: Biological: DTaP-IPV mkc vaccine

INTERVENTIONS:
Biological: DTaP-IPV vero vaccine — DTaP-IPV vero 0.5 mL solution for intramuscular injection at 2, 3½, 5 and 16 months of age
  Arms: A
Biological: DTaP-IPV mkc vaccine — DTaP-IPV mkc 0.5 ml solution for intramuscular injection at 2, 3½, 5 and 16 months of age
  Arms: B

SUMMARY:
The trial is a parallel group, multi-centre, randomized, double blind, non-inferiority trial investigating the immunogenicity and safety of two DTaP-IPV combination vaccines:

A)The investigational vaccine: DTaP-IPV containing IPV produced in a vero-cell line (DTaP-IPVvero) B)The reference vaccine: DTaP-IPV containing IPV produced in monkey kidney cells (DTaP-IPVmkc) The DTaP-IPV vaccines are administered to healthy infants at 2, 3½, 5, and 16 months of age concomitantly with Act-HIB vaccine administered as a separate injection in the opposite thigh.

Three blood samples are collected at 6, 16 and 17 months of age. Sera are analyzed for antibodies against diphtheria, tetanus, pertussis, polio and prp.

ELIGIBILITY:
Inclusion Criteria:

* The parents were informed about the trial and have signed the consent form
* The subject is healthy
* The subject has an age of 28 to 49 days at hepatitis B vaccination
* The subject had a birth weight of ≥2500 g
* The subject has received a hepatitis B vaccination at birth
* The parents grant access to the subject's medical records
* The parents are likely to comply with instructions

Exclusion Criteria:

* The subject suffers from a severe chronic disease
* The subject has already been immunized with one or more doses of diphtheria, tetanus, pertussis, poliomyelitis, or Hib vaccines
* The subject has a known allergy to one of the vaccine components or to any of the constituents of the vaccines, including Act-HIB® and hepatitis B vaccines
* The subject has a history of diphtheria, tetanus, pertussis, poliomyelitis, hepatitis B, or Hib infections
* The subject has a known congenital or acquired immunodeficiency
* The subject is in treatment with or has been in treatment with a product which is likely to modify the immune response (i.e. immunoglobulin, systemic corticosteroids, blood products, other vaccines)
* The subject is participating in another clinical trial

Ages: 28 Days to 49 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 817 (Actual)
Dates: Start 2003-09; Primary Completion 2006-10 (Actual); Study Completion 2006-10 (Actual)

PRIMARY OUTCOMES:
Simultaneous seroprotection percentages for neutralizing poliovirus antibodies (types 1, 2 and 3), when the defined limits of seroprotection is a titre value of >=4 for each of the three poliovirus types | One month after the third vaccination

CONTACTS AND LOCATIONS:
Overall Officials: Jacek Pietrzyk, Proffessor M.D., Principal Investigator — Jagellonian University, Krakow, Poland
Locations (5):
- Poland (5):
  - Centre Bydgoszcz, Bydgoszcz
  - Centre Krakow, Krakow
  - Centre Lodz, Lodz
  - Centre Poznan, Poznan
  - Centre Wroclaw, Wroclaw